CLINICAL TRIAL: NCT06857773
Title: Hepatic Arterial Infusion PUMP Chemotherapy Combined With Systemic Therapy Versus Systemic Therapy Alone as Induction Therapy for Initially Unresectable Colorectal Liver Metastases: a Randomised Controlled Trial
Brief Title: Induction Treatment for Initially Unresectable Colorectal Liver Metastases: Combined Hepatic Arterial Infusion Pump Therapy With Systemic Therapy
Acronym: PUMP-IT RCT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M23PIT; 2023-506194-35-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-01; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Neoplasms; Floxuridine; Liver Metastases; Vascular Access Device
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Floxuridine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- A: systemic therapy according to standard of care (Active Comparator): Patients included in the control arm will receive systemic therapy according to standard of care
  Interventions: Drug: Systemic therapy (standard of care)
- B: combined HAIP-therapy and systemic therapy (Experimental): Patients included in the experimental arm undergo surgery for pump placement and resection of the primary tumor. Followed by combined induction treatment with floxuridine via the hepatic arterial infusion pump (1cycle is 4 weeks) and systemic therapy (FOLFOX or FOLFIRI, 1 cycle is 2 weeks)
  Interventions: Drug: Intra arterial infusion Floxuridine (FUDR) combined with systemic therapy; Device: Hepatic arterial infusion pump (HAIP)

INTERVENTIONS:
Drug: Intra arterial infusion Floxuridine (FUDR) combined with systemic therapy — Floxuridine is administered via the hepatic arterial infusion pump directly to the hepatic artery with a continous flowrate for a period of 2 weeks. Intra arterial infusion of FUDR is combined with systemic therapy (FOLFOX/FOLFIRI) intravenously. Administration of FUDR via the chemopump is every 4 weeks and systemic therapy is administered every 2 weeks.
  Arms: B: combined HAIP-therapy and systemic therapy
Device: Hepatic arterial infusion pump (HAIP) — The HAIP (pump) is implanted during surgery combined with resection of the primary tumor before start of induction treatment with Floxuridine and concomitant systemic therapy
  Arms: B: combined HAIP-therapy and systemic therapy
Drug: Systemic therapy (standard of care) — Patient included in the control arm will receive systemic therapy according to standard clinical practice. Induction therapy regimens include: CAPOX (3 weekly) or FOLFOX/FOLFIRI/FOLFOXIRI (2weekly) with optional addition of Bevacizumab (2 weekly)
  Arms: A: systemic therapy according to standard of care

SUMMARY:
The goal of this randomized clinical trial is to investigate induction treatment with Hepatic Arterial Infusion Pump therapy combined with systemic therapy (HAIP-SYST) in chemotherapy-naive patients with unresectable colorectal liver metastases without extrahepatic disease. The main question it aims to answer is if combined HAIP-SYST improves survival compared to induction treatment with systemic therapy alone. Patients in the control arm will receive systemic therapy according to standard of care.

Study procedures experimental arm

* Surgery for pump placement and resection of the primary tumor
* Pre- and postoperative imaging (CT-anghiography, 99mTc-MAA scintigraphy)
* Induction treatment with hepatic arterial infusion pump therapy with Floxuridine combined with systemic therapy

Study procedures both arms

* Evaluation of resectability status by a National Liver Panel with surgeons and radiologists
* Questionnaires for Quality of Life

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically confirmed colorectal adenocarcinoma.
* Unresectable synchronous CRLM according to a National Liver Panel (CT-scan obtained ≤ 4 weeks prior to registration).
* No extrahepatic metastases. Patients with small (≤ 10 mm) extrahepatic lesions that are not clearly suspicious of metastases are eligible.
* No previous systemic therapy for colorectal cancer.
* Positioning of a catheter for HAIP chemotherapy is technically feasible based on imaging. The default site for the catheter insertion is the gastroduodenal artery (GDA). Accessory or aberrant hepatic arteries are no contra-indication for catheter implantation. The GDA should have at least one branch to the liver. Accessory or aberrant hepatic arteries should be ligated to allow for cross perfusion to the entire liver through intrahepatic shunts. Patients with celiac trunk stenosis are not eligible. Patients with both a replaced right and replaced left hepatic artery are not eligible.
* ECOG performance status 0 or 1.
* Life expectancy of at least 12 weeks.
* Known mutation status of RAS and BRAFV600E.
* Primary tumour in situ and resectable without neoadjuvant therapy.
* Patient is eligible for surgery.
* Patient is eligible for doublet chemotherapy.
* Laboratory requirements: i.e. adequate bone marrow, liver and renal function (obtained within 15 days prior to registration).

  * Hb ≥ 5.5 mmol/L
  * absolute neutrophil count (ANC) ≥1.5 x 109/L
  * platelets ≥100 x 109/L
  * total bilirubin ≤ 1.5 times the upper limit of normal (ULN)
  * ASAT/AST ≤ 5 x ULN
  * ALAT/ALT ≤ 5 x ULN
  * alkaline phosphatase ≤ 5 x ULN
  * Serum creatinine ≤ 1.5 x upper limit of normal or a MDRD (eGFR) ≥ 45 ml/min;
  * Prothrombin time or INR < 1.5 x ULN, unless coumarin derivates are used. All patients using coumarin derivates will be treated with LMWH or DOAC instead.
* Before registration, written informed consent must be given and signed according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Prior hepatic radiation, resection, or ablation.
* Any malignancy, comorbidity or condition that interferes with the planned study treatment or the prognosis of CRLM, determined by the treating physician.
* History of prior malignancy except for the following: (a) malignancy treated with curative intent and with no evidence of active disease present within 3 years prior to inclusion, (b) curatively treated malignancies felt to be at low risk for recurrence by treating physician and MDT, (c) adequately controlled nonmelanomatous skin cancer, (d) adequately treated carcinoma in situ without current evidence of disease.
* Obstructive primary tumour requiring emergency surgery, primary tumour necessitating a multivisceral resection/abdominoperineal resection or a rectal tumour requiring preoperative short-course radiotherapy or chemoradiotherapy for local tumour control.
* MMR deficiency.
* DPD-deficiency.
* Pregnant or lactating women.
* Serious concomitant systemic disorders that would compromise the safety of the patient or his/her ability to complete the study, at the discretion of the investigator.
* Organ allografts requiring immunosuppressive therapy.
* Serious non-healing wound, ulcer, or bone fracture.
* Chronic treatment with corticosteroids (dose of ≥ 10 mg/day methylprednisolone equivalent excluding inhaled steroids).
* Known serious infections (uncontrolled or requiring treatment).
* History of psychiatric disability judged by the investigator to be clinically significant, precluding informed consent or interfering with compliance for HAIP-SYST or standard systemic therapy.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
* Underlying liver disease including liver fibrosis and cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to five years after randomization
  Defined as the time between randomization and the event of death.

SECONDARY OUTCOMES:
Progression-free survival | Up to five years after randomization
  Defined as the time between randomization and the first event defined as recurrence or death, whichever comes first.
Hepatic progression-free survival | Up to five years after randomization
  Defined as the time between randomization and the event of progression confined to the liver.
Conversion to resection rate | if CRLM convert to resectable, often at 3-6 months after start induction treatment
  Defined as conversion surgery with intention of complete local treatment of all CRLM
Complete local treatment rate | if CRLM convert to resectable, often at 3-6 months after start induction treatment
  R0/1 resection or ablation of all visible CRLM
Objective response rate (ORR) | During protocol treatment, up to 6 months of induction treatment
  Defined as complete or partial response according to RECIST 1.1
Disease control rate (DCR) | During protocol treatment, up to 6 months of induction treatment
  Defined as a complete or partial and stable disease
Pathological response rate | Pathological assessment of conversion surgery after induction treatment
  Defined as a major and complete pathological response of resected lesions according to the Mandard score.
Surgical complication rate | at 30 days an 90 days postoperatively
  of HAIP placement and/or any tumour related surgery. Defined as the percentage of surgery-related (HAIP placement and/or any protocol tumor related surgery) complications grade ≥3 according to the Clavien-Dindo classification
Adverse events and toxicity of HAIP-SYST and systemic therapy | During protocol treatment
  Defined as the percentage of treatment related AEs grade ≥ 3 according to Common Terminology Criteria for Adverse Events (CTCAE), version 5.0
Quality of Life (QoL) | Up to five years after randomization
  Assessed by standardized Quality of Life questionnaires (EORTC QLQ-C30 & EQ-5D3L)
Cost-effectiveness | Up to five years after randomization
  Expressed by costs per quality adjusted life years (QALYs) and estimated according to the Health Technology Assessment (HTA) methods. Productivity loss is assessed by adjusted standardized Productivity Costs Questionnaires (iPCQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Antoni van Leeuwenhoek-Netherland Cancer Institute, Amsterdam, Netherlands